CLINICAL TRIAL: NCT02357238
Title: Genetics of Uveitis
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Sunil Srivastava, Staff physician, The Cleveland Clinic
Other Study IDs: 11-087
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Uveitis; Infectious Uveitis
Keywords: Uveitis; Infectious
MeSH Terms: conditions — Uveitis; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole blood serum will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Uveitis: Uveitis or infectious uveitis patients

SUMMARY:
In order to improve the investigators knowledge about uveitis and the underlying mechanism of disease, the investigators propose collecting blood from patients with uveitis, isolating DNA and sequencing the DNA to identify genetic mutations or associations in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient above with the diagnosis of uveitis.
* Any patient with a diagnosis of infectious uveitis such as toxoplasmosis retinochoroiditis, herpes associated retinitis.

Exclusion Criteria:

* Patients who are unable to give consent
* Patients in whom an adequated blood sample can not be obtained.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient able to sign an informed consent or child of age 6 with parental /guardian consent with the diagnosis of uveitis or infectious uveitis.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Non infectious uveitis | 5 years
  Distinct uveitis conditions will have a polymorphism association or specific mutation.

SECONDARY OUTCOMES:
Infectious uveitis | 5 years
  Infectious uveitis (such as herpes associated uveitis, toxoplasmosis retinochoroiditis) will have specific polymorphisms/mutations in innate immune system genes which predispose the patient to infectious uveitis.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil K. Srivastava, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No